CLINICAL TRIAL: NCT02397421
Title: Research Into the Effect of SGLT2 Inhibition on Left Ventricular Remodeling in Patients With Heart Failure and Diabetes Mellitus
Brief Title: Safety and Effectiveness of SGLT-2 Inhibitors in Patients With Heart Failure and Diabetes
Acronym: REFORM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Principal Investigator, Jagdeep Singh Surmukh Singh, Dr, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-002742-42
Record Dates: First submitted 2015-03-12; First posted 2015-03-25 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure; Diabetes
Keywords: Heart failure; Diabetes; Left ventricular remodelling; SGLT-2 inhibitors
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Dapagliflozin 10mg once daily
  Interventions: Drug: Dapagliflozin
- Control (Placebo Comparator): Capsules containing microcrystalline cellulose Ph Eur overencapsulated in a hard gelatine capsule shell to match the active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Sodium Glucose Linked Transporter Type 2 (SGLT-2) Inhibitor
  Other Names: Forxiga
  Arms: Treatment
Drug: Placebo — Capsules containing microcrystalline cellulose Ph Eur overencapsulated in a hard gelatine capsule shell to match the active comparator
  Arms: Control

SUMMARY:
Patients with diabetes are at increased risk of developing heart failure (HF) which can lead to increased shortness of breath, reduced ability to exercise and in some cases premature death as the heart becomes less efficient at pumping blood around the body. However the treatment options for such patients remain limited.

This study will test the safety and benefits of using a new class of drug, the SGLT2 Inhibitor (Dapagliflozin), in treating HF and diabetes.

Participants will have a Magnetic Resonance Imaging (MRI) scan of the heart, to measure the efficiency and the extent of thickening of the heart muscle before they start on treatment of dapagliflozin, or placebo for one year. They will also do exercise testing on an exercise bike (if capable) and a walking test plus fill in some questionnaires on how their heart failure affects their quality of life. Participants will then continue as normal with currently prescribed medication for their diabetes and heart failure. After a year the tests will be repeated to determine if patients receiving Dapagliflozin benefited more than those who weren't on the drug.

This study is funded by the European Foundation for the Study of Diabetes (EFSD)

DETAILED DESCRIPTION:
Men and women with diabetes have a 2-5-fold increased risk of heart failure (HF). The prevalence and incidence of HF is increasing in diabetes and mortality rates remain alarmingly high. This highlights the need for novel therapies in diabetes that will reduce HF risk and /or delay disease progression.

Drug options are currently limited as some diabetic therapies such as thiazolidinediones are contra-indicated in HF. SGLT2 inhibitors, the newest class of anti-diabetic drugs, are an exciting new approach to diabetes management that may have additional beneficial effects in diabetes and HF. SGLT2 inhibitors may have beneficial effects on adverse left ventricular (LV) remodelling that occurs in patients with diabetes and heart failure by reducing the load on the heart through its diuretic and blood pressure lowering actions.

Exercise intolerance is a cardinal symptom of patients with HF and improving insulin sensitivity has been shown to improve exercise capacity. SGLT2 inhibition has been shown to improve insulin sensitivity and to reduce weight and therefore has the potential to improve exercise capacity in HF.

This study will assess the potential beneficial effects of the oral SGLT2 inhibitor, dapagliflozin, on LV remodelling and exercise capacity in patients with diabetes and HF. The findings of this study may help to establish the utility of SGLT2 inhibitors in diabetic patients with HF and provide important clinical data on the impact of SGLT2 inhibition on LV remodelling.

ELIGIBILITY:
Inclusion Criteria:

* were previously diagnosed with Type 2 Diabetes
* are diagnosed with NYHA functional class I-III HF with prior echocardiographic evidence of Left Ventricular Systolic Dysfunction (LVSD) (At least mild LV systolic dysfunction on sonographer assessment or ejection fraction at 45% or less)
* on furosemide 80mg daily or less, or equivalent loop diuretic
* have stable HF symptoms for at least three months prior to consent
* on stable therapy for HF for at least three months prior to consent
* have not been hospitalised for HF for at least three months prior to consent

Exclusion Criteria:

* severe hepatic disease
* renal disease defined as Chronic Kidney Disease (CKD) class 3b or worse (i.e. estimated glomerular filtration rate (eGFR) / creatinine clearance CrCl <45ml/min)
* systolic BP <95mmHg at screening visit
* screening HbA1c <6.0%
* unable to walk to perform cardio pulmonary exercise testing or 6MWT
* malignancy (receiving active treatment) or other life threatening diseases
* pregnant or lactating women
* any contraindication to MRI (e.g. claustrophobia, metal implants, penetrative eye injury or exposure to metal fragments in eye requiring medical attention)
* patients who have participated in any other clinical trial of an investigational medicinal product within the previous 30 days
* patients who are unable to give informed consent
* any other reason considered by a study physician to be inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in LV end systolic volume (absolute value and indexed for BSA) or LV end diastolic volume (absolute value and indexed for BSA) | 1 year
  Cardiac MRI will be performed to determine the change in end systolic and diastolic volumes between both groups of patients

SECONDARY OUTCOMES:
Change in LV mass, LV ejection fraction, RV end diastolic volume, RV end systolic volume, RV ejection fraction, atrial dimensions and volumes, and LV remodelling index (LV mass / LVEDV) | 1 year
  MRI will be performed to study the effects of the intervention on various other cardiac parameters.
Fluid status (Bioelectrical Impedence Analysis (BIA) | 1 year
  Bioelectrical Impedence Analysis (BIA) will be conducted to determine the effect of the study dug on overall fluid balance
Objective functional capacity (6 Minute Walk Test (6MWT) | 1 year
  6 Minute Walk Test (6MWT) will be performed to objectively determine the functional capacity of participants
Exercise capacity (Cardio-pulmonary Exercise Testing (CPET) | 1 year
  Cardio-pulmonary Exercise Testing (CPET) will be performed to determine the exercise capacity of participants
Quality of life (Minnesota Living with Heart Failure and SF-36 questionnaire) | 1 year
  will be conducted to determine the impact of the intervention on subjective quality of life
Cardiac and inflammatory biomarkers | 1 year
  Brain natriuretic peptide (BNP) and other inflammatory & oxidative stress markers will be measured
Diuretic requirement (total diuretic requirement to maintain euvolemia) | 1 year
  The total diuretic requirement to maintain euvolemia will be compared between the beginning and end of the trial
Change in degree of microalbuminuria | 1 year
  Urinary analysis will be performed to determine if there has been any change in the severity of microalbuminuria
Quantify amount of natriuresis | 1 year
  Urinary analysis will be performed to quantify the amount of sodium excretion.
The safety of dapagliflozin use in diabetic, heart failure patients with regard to worsening HF, hospitalization and death will be evaluated | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jagdeep Singh, MBBS, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital and Medical School, Dundee, Angus, United Kingdom

REFERENCES:
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515
- [Derived] Singh JSS, Mordi IR, Vickneson K, Fathi A, Donnan PT, Mohan M, Choy AMJ, Gandy S, George J, Khan F, Pearson ER, Houston JG, Struthers AD, Lang CC. Dapagliflozin Versus Placebo on Left Ventricular Remodeling in Patients With Diabetes and Heart Failure: The REFORM Trial. Diabetes Care. 2020 Jun;43(6):1356-1359. doi: 10.2337/dc19-2187. Epub 2020 Apr 3. PMID 32245746
- [Derived] Singh JS, Fathi A, Vickneson K, Mordi I, Mohan M, Houston JG, Pearson ER, Struthers AD, Lang CC. Research into the effect Of SGLT2 inhibition on left ventricular remodelling in patients with heart failure and diabetes mellitus (REFORM) trial rationale and design. Cardiovasc Diabetol. 2016 Jul 15;15:97. doi: 10.1186/s12933-016-0419-0. PMID 27422625